CLINICAL TRIAL: NCT01487122
Title: Microwave Diathermy for Treating Nonspecific Chronic Neck Pain. A Randomised Controlled Trial
Brief Title: Microwave Diathermy for Treating Nonspecific Chronic Neck Pain
Acronym: MOFIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Health Service of Andalucia (Other Government)
Responsible Party: Principal Investigator, Juan Alfonso Andrade Ortega, Head of Physical Medicine and Rehabilitation, Health Service of Andalucia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MOjaao
Record Dates: First submitted 2011-12-01; First posted 2011-12-07 (Estimated); Last update posted 2011-12-07 (Estimated); Status verified 2011-12

CONDITIONS: Neck Pain
Keywords: Diathermy; Neck Pain
MeSH Terms: conditions — Neck Pain; Fever

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Continuous Microwave (Experimental)
  Interventions: Radiation: Continuous microwave
- Pulsed Microwaves (Experimental)
  Interventions: Radiation: Pulsed microwaves
- sham microwaves (Sham Comparator)
  Interventions: Procedure: Sham microwaves

INTERVENTIONS:
Radiation: Continuous microwave — Continuous microwave through a great circular electrode, 15 cm from the neck, 20 minutes, 80 watts, 15 sessions in 3 weeks
  Arms: Continuous Microwave
Radiation: Pulsed microwaves — Pulsed microwaves through a great circular electrode, 15 cm away from the neck, 20 minutes, 80 watts, 15 sessions in 3 weeks
  Arms: Pulsed Microwaves
Procedure: Sham microwaves — Unplugged microwave generator, great circular electrode, 15 cm away from the neck, 20 minutes, 15 sessions in 3 weeks
  Arms: sham microwaves

SUMMARY:
This randomised controlled trial aims to compare the effect of microwave diathermy (continuous and pulsed modes) with sham microwave diathermy in nonspecific chronic neck pain patients. Every patient will also be treated by exercise and transcutaneous electrical neurostimulation (TENS). The primary endpoint is to establish whether the use of microwaves is justified in terms of pain relief or reduction of disability in this patients.

ELIGIBILITY:
Inclusion Criteria:

* to be between 18 and 65 years old
* to be diagnosed with chronic nonspecific neck pain (i.e. during more than 3 months in the absence of red flags (unexplained weight loss, fever, neurological signs, history of cancer, history of inflammatory conditions...)

Exclusion Criteria:

* pregnancy
* sick leave
* litigation
* claims because the neck pain.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2008-09; Primary Completion 2011-06 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in pain at six months | Baseline. At three weeks. At six months
  Pain as measured by visual analogic scale
Change from baseline in neck disability at six months | Baseline. At three weeks. At six months
  Neck disability as measured by "Neck Disability Index" and "Northwick Park Neck Pain Questionnaire"
Change from baseline in quality of life at six months | Baseline. At three weeks. At six months
  Quality of life as measured by SF-36 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Juan A Andrade Ortega, MD, Principal Investigator